| 1<br>2 | Hybrid Closed Loop Therapy and Verapamil for Beta Cell Preservation in New Onset<br>Type 1 Diabetes: |
|---|---|
| 3 | A Proof-of-Concept Study |
| 4 | |
| 5 | Statistical Analysis Plan |
| 6 | Version 2.0 |
| 7 | |
| 8 | Corresponds to Version 5.2 of the protocol |
| 9 | |
| 10 | |
| 11 | |
| 12 | |
| 13 | |
| 14 | |
| 15 | |
| 16 | |
| 17 | |
| 18 | |
| 19 | |
| 20 | |
| 21 | |
| 22 | |
| 23 | |
| 24 | |
| 25<br>26 | |
| 20<br>27 | |
| <u>-</u> / | |

# 28 Version History

| SAP<br>Version | Author | Approver | Effective<br>Date | Revision<br>Description | Study Stage | Protocol<br>Version |
|---|---|---|---|---|---|---|
| 1.0 | Rob<br>Henderson<br>& Colleen<br>Bauza | Craig<br>Kollman | 07May2020 | Original Version | Enrollment has not started yet | 4.1 |
| 1.1 | Colleen<br>Bauza | Craig<br>Kollman | 17 Feb2021 | Added conditions to calculate c-peptide; corrected typos | Enrollment ongoing | 4.4 |
| 1.2 | Colleen<br>Bauza | Craig<br>Kollman | 20 April<br>2021 | Added condition to HCL per-protocol analysis | Enrollment ongoing | 4.4 |
| 1.3 | Ryan<br>Bailey | Craig<br>Kollman | 14 July<br>2022 | Revised methods for handling skewed outcomes | Enrollment completed. Follow-up ongoing | 5.2 |
| 2.0 | Ryan<br>Bailey | Craig<br>Kollman | 27<br>September<br>2022 | Included type of device as a fixed effect in models comparing CGM metrics between verapamil and placebo groups. Added more subgroup analyses. Replaced hospitalizations with SAEs as a safety metric. | Enrollment completed.<br>Follow-up ongoing | 5.2 |

Ryan Bailey I am digitally signing this document 2022-09-27 14:14-04:00 30 31 Author: \_ 32 Craig Kollman 33 I am digitally signing this document 2022-09-27 14:45-04:00 34 Senior Statistician: \_\_ 35 Colleen Bauza 36 I am digitally signing this document 2022-09-28 15:38-04:00 JCHR Project Director: \_ 37

38

| 39 | Digitally signed by Gregory P. Gregory P. Forlenza Forlenza |
|---|---|
| 40 | Protocol Co-Chair |
| 41 | |
| 42 | MutainAt Man. 30et 2002 |
| 43 | Protocol Co-Chair The Control of the |
| 44 | · · |
| 45 | |

# 1. Study Overview

- 47 The purposes of this study are to
  - 1) to determine if initiation of HCL therapy plus intensive diabetes management soon after diagnosis of stage 3 T1D can achieve near-normalization of glucose concentrations that preserves beta cell function (Cohort A and Cohort B will be combined for the analysis)
  - 2) to determine if oral verapamil started soon after diagnosis of stage 3 T1D preserves beta cell function (Cohort A)

- There are two cohorts in this trial
  - A) body weight ≥30 kg
  - B) body weight <30 kg

- Randomization schedules will be separate for Cohort A and Cohort B and will be stratified by site. Cohort A will be participating in a factorial design arm. Eligible participants will be randomly assigned (1:1:1:1) to one of 4 groups:
  - HCL and placebo
  - HCL and verapamil
  - non-HCL and placebo
  - non-HCL and verapamil.

Cohort B will be not be assigned to verapamil due to their lower body weight. These participants will be randomly assigned 2:1 to either HCL or non-HCL.

Participants assigned to HCL will receive intensive diabetes management with frequent contacts by study staff with the goal of near-normalization of glucose concentrations. Participants assigned to non-HCL will receive a Dexcom G6 CGM and diabetes management will follow usual care.

Participants will be followed for 12 months from diagnosis, with visits timed from diagnosis at 6, 13, 26, 39, and 52 weeks. Participants will have a mixed meal tolerance test (MMTT) performed, HbA1c measured, insulin dose (units/kg/day) recorded, CGM data uploaded, and pregnancy testing performed (if indicated) at some or all of the previously noted timepoints.

- Additional Procedures for Cohort A
- Drug will be double blinded. Cohort A will have additional safety visits 1 week after initiation of study drug and after each study drug dose increase.

# 2. Consistency of Statistical Analysis Plan with Protocol

- Prior to the start of the study, the following secondary outcomes have been added that were not specified in the protocol:
  - Percentage of participants with peak C-peptide ≥ 0.2 pmol/ml
  - Percentage of time sensor glucose from 70 to 140 mg/dL
  - Percentage of participants with ≥70% of sensor glucose values from 70 to 180 mg/dL
  - Percentage of time sensor glucose > 140 mg/dL
    - Total daily insulin per kg
    - Basal: Bolus ratio

92 93

84

87

88

89

90

91

- 94 Serious adverse events has been added as a safety outcome in place of hospitalizations.
- Otherwise, the author of this SAP has verified that the analyses described in this document are consistent with the version of the protocol listed in the version history table above.

97 98

# 3. Primary Statistical Hypotheses

The primary outcome is the C-peptide area under the curve (AUC) in response to a 2-hour MMTT at 52 weeks.

100101102

103

104

105

106

107

99

#### 3.1 HCL vs. non-HCL

- *Null Hypothesis*: There is no difference in the C-peptide AUC in response to a 2-hour MMTT at 52 weeks between HCL with intensive care and non-HCL with standard care for the combined Cohort A and B population.
- Alternative Hypothesis: There is a nonzero difference in the C-peptide AUC in response to a 2-hour MMTT at 52 weeks between HCL with intensive care and non-HCL with standard care for the combined Cohort A and Cohort B population.

108109110

111

112

113

114

### 3.2 Verapamil vs. Placebo

- *Null Hypothesis:* There is no difference in the C-peptide AUC in response to a 2-hour MMTT at 52 weeks between verapamil and placebo for the Cohort A population.
- Alternative Hypothesis: There is a nonzero difference in the C-peptide AUC in response to a 2-hour MMTT at 52 weeks between verapamil and placebo for the Cohort A population.

115116

117

### 4. Sample size

- 118 The sample size calculation is detailed in a separate document and is summarized below. Sample
- size was driven by the verapamil vs. placebo comparison as the test only includes participants in
- 120 Cohort A. The mean of the transformed C-peptide (log(AUC + 1)) and the root mean square
- error in the placebo group were assumed to be 0.315 and 0.18, respectively, based on 90% CIs
- from prior studies (1). The corresponding geometric-like mean C-peptide value of 0.370
- pmol/mL was calculated using the inverse transformation:  $\exp(0.315) 1$ . A recent randomized
- trial (2) found a 62% increase in mean C-peptide in verapamil compared with placebo, although

- the total sample size was small (N=24) and confidence intervals were wide. Therefore, this
- study assumed a smaller, 50% increase in mean C-peptide using verapamil. The expected
- geometric-like mean C-peptide value in the verapamil arm was  $0.370 \cdot 1.50 = 0.555$  pmol/mL.
- After a log(x+1) transformation, the mean values in the control and treatment groups are 0.315
- and 0.441, respectively, giving a treatment effect of 0.441-0.315=0.126.
- With these estimates, a sample size of 88 participants in Cohort A was calculated to provide 90%
- power with a 5% two-sided type 1 error rate and a 1:1 treatment group allocation to detect a
- verapamil vs. placebo treatment group difference assuming the true relative difference between
- groups was 50%. To account for a 10% dropout rate, the sample size in Cohort A will be 98
- participants.
- A sample size of 33 participants for Cohort B was selected based on convenience. Participants
- in Cohort B will be allocated to either HCL or non-HCL in a 2:1 treatment group allocation.
- Thus, 131 participants are expected tobe enrolled in either Cohort A or Cohort B with
- approximately 71 participants in HCL/intensive care and 60 participants in non-HCL/standard
- care arm. Assuming around a 10% dropout rate, an HCL/intensive care treatment effect of 50%,
- and an upper confidence limit estimate of 0.18 for the standard deviation (same presumed
- estimates for verapamil vs. placebo comparison), this study has 96% power to detect a significant
- HCL/intensive care vs. non-HCL/standard care treatment group difference with a type 1 error
- 143 rate of 5%.

#### 5. Outcome Measures

- 146 Primary Efficacy Outcome
- 147 The primary outcome is the C-peptide in response to a 2-hour MMTT at 52 weeks. This is
- measured as the area under the stimulated C-peptide curve (AUC).

149

152

153

- 150 <u>Secondary Efficacy Outcomes</u>
- 151 *C-peptide* 
  - C-peptide AUC at 13, 26, and 39 weeks (52 weeks is primary outcome)
  - Peak C-peptide during a 2-hour MMTT at 13, 26, 39, and 52 weeks
- Percentage of patients with peak C-peptide  $\geq 0.2$  pmol/ml at 13, 26, 39, and 52 weeks

155

- 156 CGM Metrics
- 157 The following CGM-derived indices will be computed over the study period for 24 hours,
- daytime (6:00am to 11:59pm) and nighttime (midnight to 5:59am) at 6, 13, 26, 39, and 52 weeks:
- Mean glucose
  - Percentage of time sensor glucose from 70 to 180 mg/dL
- Percentage of time sensor glucose from 70 to 140 mg/dL
- Percentage of patients with ≥70% of sensor glucose values from 70 to 180 mg/dL
- Percentage of time sensor glucose >140 mg/dL
- Percentage of time sensor glucose >180 and >250 mg/dL

- Percentage of time sensor glucose <54 and <70 mg/dL</li>
  Coefficient of variation
  HbA1c
  Values at 13, 26, 39, and 52 weeks will include the following:
- Mean HbA1c

• Percentage of patients with an HbA1c <7.0% and <6.5%

173 Insulin

- 174 Values at 6, 13, 26, 39, and 52 weeks
  - Total daily insulin per kg
  - Basal: Bolus ratio

176 177 178

181

175

171172

# 5.1 C-Peptide

### 179 Area Under the Curve (AUC)

The stimulated C-peptide AUC will be calculated for an MMTT if the following conditions hold:

- A C-peptide measurement available at 0 minutes.
- At least three C-peptide measurements available among the following 5 times: 15 minutes, 30 minutes, 60 minutes, 90 minutes, and 120 minutes.
  - At least one C-peptide measurement available at 90 minutes or 120 minutes.
  - No two consecutive C-peptide measurements missing.

185 186 187

188

189

184

If any of these conditions is violated, the C-peptide AUC will be treated as a missing value for that visit. If it is discovered that the MMTT was completed while the participant was in closed loop or while the participant was not fasting, those MMTT results will also be treated as missing for that visit.

190 191

192 If the lab deems the C-peptide AUC value to be below the lower limit of detection (LLOD), the C-peptide value will be assigned the value of ½ of the LLOD, akin to TrialNet (3).

194 195

For each MMTT, the starting time of the MMTT will be defined as t=0 if the C-peptide value is available at that time point.

196 197 198

199

The trapezoidal rule will be used to calculate the stimulated C-peptide AUC as a weighted sum of the C-peptide measurements. Throughout the calculation, target times for C-peptide measurements will be used (as opposed to the actual measurement times).

200201202

203

204

205

If the C-peptide measurement at 120 minutes is not available, the following steps will be used to calculate AUC:

- Calculate AUC<sub>90</sub> from C-peptide measurements taken between baseline and 90 minutes
- Calculate AUC as AUC<sub>90</sub> × (120/90)

206

### 207 *Peak*

- This will be defined as the maximum of all C-peptide values during the MMTT, which can occur
- 209 at t=0. The rules for handling any missing measurements during the MMTT will be the same as
- 210 listed above for the AUC. Thus, peak C-peptide will be missing for a visit if and only if C-
- 211 peptide AUC is also missing.

### 212 5.2 CGM Metrics

- Note that no pre-randomization CGM data are collected in this protocol (new onset patients) so no
- baseline CGM metrics will be calculated.

215

- Participants assigned to a non-HCL group will be provided a commercially available Dexcom G6
- 217 CGM. Participants who stop using a CGM or have insufficient CGM data will wear a blinded
- Dexcom G6 for approximately 10 days at 6, 13, 26, 39 and 52 weeks. The CGM indices listed
- above will be computed separately at each follow-up visit including all unblinded data 28 days
- prior to the visit date and any data from a blinded sensor placed at the visit (or prior to the visit at
- 52 weeks). A minimum of 5 days (120 hours) of CGM data will be required to calculate CGM
- 222 indices at each visit.

223

- For daytime (6:00am to 11:59pm) versions of the CGM metrics, at least 80 hours of data will be
- required; and for the nighttime versions (midnight to 5:59am), at least 40 hours of data will be
- 226 required.

227 228

# 6. Primary Analyses

- 229 Primary analyses will follow the intent to treat principle. Primary outcome is C-peptide AUC at
- the 52-week visit. The protocol window is 52-weeks from diagnosis  $\pm$  14 days, but out-of-
- window MMTT results will be included in the analysis if obtained within 52 weeks from
- diagnosis  $\pm$  42 days (Day 322-406 from the date of diagnosis). Any MMTT results outside this
- analysis window will be excluded from the primary analysis and treated as missing data.

234

235

### 6.1 HCL vs. non-HCL

- The HCL/intensive care versus non-HCL/standard care comparison will combine participants from
- 237 Cohort A and B. Comparisons for HCL versus non-HCL will be pooled over verapamil groups
- 238 (verapamil, placebo, neither [Cohort B]). Summary statistics appropriate to the distribution, mean
- (SD) or median (quartiles) of log(AUC+1), will be tabulated for each treatment group at 52 weeks.
- Boxplots, with HCL vs Non-HCL groups next to each other, will be produced for each visit.

- 242 A constrained longitudinal regression model will be constructed with log(AUC+1) as the
- 243 dependent variable controlling for age, time from diagnosis to randomization, verapamil group
- 244 (verapamil, placebo, or neither [Cohort B]), and clinical site (random effect). C-peptide values at
- baseline, 13, 26, 39 and 52 weeks will be included in the longitudinal model which will account
- for the correlated data from the same participant using an unstructured covariance matrix. If there
- 247 are convergence issues, a simpler covariance structure (e.g., autoregressive or compound

symmetry structure) will be used. The model specified above is equivalent to adjusting for baseline as a covariate, but also has the advantage of being able to handle any cases of missing baseline.

250251

252

A time by treatment (HCL) interaction will be included in the model so that different treatment effects can be estimated. The treatment effect at 52 weeks from this model (point estimate, 95% confidence interval (CI), and p-value) will be reported as the primary analysis results.

253254

The log(AUC+1) transform is expected to make the residuals normally distributed, but regression diagnostics will be performed to check the residuals. If the residuals have a skewed distribution then robust regression using M-estimation will be used.

258

259 Missing data will be handled by the method of direct likelihood.

260

261

### 6.2 Verapamil vs. Placebo

The verapamil vs. placebo comparison will only include participants in Cohort A and will be pooled over the HCL and usual care groups.

264

Summary statistics appropriate to the distribution, mean (SD) or median (quartiles) of log(AUC+1), will be tabulated for verapamil versus placebo at 52 weeks.

267

A similar constrained longitudinal analysis will be performed controlling for HCL or no HCL as a covariate.

270 271

272

### 7. Analysis Cohorts

#### 7.1 Intent to Treat

- 273 The primary analyses will follow the intention-to-treat principle. They will include all
- 274 randomized participants, and data will be analyzed based on the treatment assigned from
- 275 randomization regardless of the actual treatment received. Unless specified, all analyses will be
- 276 ITT. As noted above, any data from an MMTT where it is known that the participant was in
- 277 closed loop at the time or the participant was not fasting will be excluded from analysis.

278279

### 7.2 Per Protocol Analyses

- In addition to ITT, per-protocol analyses for the primary outcome will be conducted for the
- 281 HCL/intensive therapy group vs. non-HCL/standard care comparison and, separately, for the
- verapamil vs. placebo comparison. The per-protocol analysis will be limited to those with non-
- 283 missing 52-week visit data.

- The per-protocol analysis for HCL/intensive therapy vs. non-HCL/standard therapy will include
- 286 HCL participants who use the HCL system at least 85% of the time over the course of the study
- and all non-HCL participants. If it is discovered that a non-HCL participant was using closed
- loop during the study, his/her data will be excluded from this per-protocol analysis.

- The per-protocol analysis for verapamil vs. placebo will only include participants in Cohort A who have taken at least 80% of the study drug (both active and placebo groups) over the course
- 292 of the study.

293

For each analysis noted above, the per-protocol analysis will not be conducted if the N for the analysis is  $\geq 95\%$  of the N in the primary intent-to-treat analysis.

296

297

### 8. Secondary Analyses

As described above for the primary analysis, comparisons of HCL versus non-HCL will include cohorts A and B and will be pooled over verapamil groups. Comparisons of verapamil versus placebo will be limited to Cohort A and will be pooled over HCL and usual care groups.

301 302

303

304

305

Descriptive summary statistics appropriate to the distribution will be given for each secondary efficacy outcome listed above in Section 5 by treatment group at each visit. Corresponding boxplot figures of baseline and 52 weeks, boxplot figures over time, scatterplots of baseline versus 52 weeks, and histograms of baseline, 26 weeks, and 52 weeks will be constructed for selected metrics.

306 307 308

### 8.1 Formal Statistical Comparisons of Treatment Groups

309 310

### C-peptide Related Secondary Efficacy Outcome

Formal statistical comparisons of treatment groups will limited to C-peptide AUC at 13, 26, and 39 weeks (52 weeks is the primary analysis described above).

312 313 314

315

316

317

318

319

320

321

322

323

324

325

311

### Other Secondary Efficacy Outcomes

- Formal statistical comparisons of treatment groups for other secondary efficacy outcomes will be limited to the following at 26 and 52 weeks:
  - Mean HbA1c
    - Total daily insulin per kg
    - Selected overall (24 hours) CGM indices:
      - > Mean glucose
      - > Percentage of time sensor glucose from 70 to 140 mg/dL
      - > Percentage of time sensor glucose from 70 to 180 mg/dL
      - > Percentage of time sensor glucose >180 mg/dL
      - > Percentage of time sensor glucose >250 mg/dL
      - > Percentage of time sensor glucose <54 mg/dL
      - > Percentage of time sensor glucose <70 mg/dL

- Separate comparisons for HCL versus non-HCL and verapamil versus placebo will be done similarly as described above for the primary analysis. Except where noted otherwise below in
- similarly as described above for the primary analysis. Except where noted otherwise below in Sections 8.3 and 8.5, the general approach for analysis of secondary outcomes will be as follows:
- For each outcome, a constrained longitudinal model will be fit adjusting for age, time from
- diagnosis to randomization, verapamil group (for HCL analysis), HCL group (for verapamil

analysis) and clinical site as a random effect. A treatment by time interaction will be included in the model and treatment effects (and 95% CI) will be reported separately at 26 and 52 weeks. Regression diagnostics and remedy for a non-normal distribution will be as described above for the primary analysis. Missing data will be handled by the method of direct likelihood.

### 8.2 Included Data

The following analysis windows will be applied to determine which data values collected at a follow-up visit will be included in the analysis. The windows indicated in the protocol are expanded here so that data collected at some out of window visits may still be included. If there are multiple visits with non-missing data values in the same analysis window, the one closest to the target date (center of window) will be used for analysis.

These windows apply to C-peptide, HbA1c, and insulin. These do not apply to the CGM metrics (see Section 5.2).

| Visit | Protocol Target Window Range a | Protocol Allowable<br>Window Range <sup>a</sup> | Proposed Analysis<br>Window <sup>a</sup> |
|---|---|---|---|
| Week 13 (3 mo) <sup>b</sup> | $91 \pm 3 \text{ days}$ | 91 ± 7 days | $91 \pm 28 \text{ days}$ |
| Week 26 (6 mo) <sup>b</sup> | $182 \pm 7 \text{ days}$ | $182 \pm 14 \text{ days}$ | $182 \pm 28 \text{ days}$ |
| Week 39 (9 mo) <sup>b</sup> | $273 \pm 7 \text{ days}$ | $273 \pm 14 \text{ days}$ | $273 \pm 28 \text{ days}$ |
| Week 52 (12 mo) <sup>b</sup> | $364 \pm 7 \text{ days}$ | $364 \pm 14 \text{ days}$ | $364 \pm 42 \text{ days}$ |

a - Days from diagnosis.

#### 8.3 C-peptide Values

The same log(x+1) transformation mentioned above for AUC values in the primary analysis will be used for both AUC and peak at all time points. Note that TrialNet refers to the back-transform of the mean of the log(x+1) values as the "geometric-like" mean. Treatment group comparisons of C-peptide AUC at 13, 26, and 39 weeks will be taken from the same longitudinal model described above for the primary analysis.

### 8.4 HbA1c

Analyses will utilize values from the central laboratory. Local HbA1c values will not be utilized.

#### 8.5 CGM Metrics

The descriptive analyses described above will be done for each CGM index listed in Section 5, separately for:

- Overall CGM data (24 hours per day)
- Daytime (limited to CGM readings from 6:00 am 11:59 pm)
- Nighttime (limited to CGM readings from midnight 5:59 am).

Boxplots and scatterplots will be limited to selected CGM metrics at each of the 3 times of the day listed above.

b - Applies to C-peptide (AUC and peak), HbA1c, and insulin.

- Formal statistical comparisons of treatment groups will be done for the selected CGM indices listed above and will be limited to the 24 hour versions (analysis of daytime and nighttime versions will be descriptive only). Analysis will follow the method described above with three exceptions:
  - The longitudinal model will not be constrained because no baseline values will be available.
  - The unconstrained longitudinal model will include 6 week values.
  - For verapamil vs. placebo comparisons the type of CGM sensor used (Medtronic, Dexcom) will be included as a covariate in the models. This covariate will be allowed to differ within subject if the participant changes devices between visits. If the participant switches sensors in the 28 day period used to calculate CGM metrics, data from both sensors will be used to calculate metrics and the value for the sensor covariate will be set equal to the sensor which contributed the most data.

It is likely that percentage of sensor values below 54 mg/dL and possible that the percentage of sensor values above 250 mg/dL will have a skewed distribution. The other CGM metrics are anticipated to have an approximate normal distribution. As described above for the primary analysis, robust regression with M-estimation will be used to analyze skewed outcomes.

The percentage of patients with ≥70% of sensor values from 70 to 140 mg/dL will be analyzed using generalized estimating equations (GEE) logistic regressions adjusting for baseline HbA1c, age, time from diagnosis to randomization. Clinical site will be treated as a repeated factor using a compound symmetry covariance structure. A risk-adjusted difference and 95% confidence interval for the percentages will be calculated using the method of Kleinman and Norton (4). This analysis will be available cases only. There will be no imputation of missing data.

### 9. Interaction Analyses

- A factorial design is being used for this study because it is believed to be unlikely that the device (HCL) and drug (verapamil) would interact with each other. An interaction test will be conducted to explore this assumption. This analysis will be limited to cohort A. Note that this study has not been powered to detect interaction. Thus, this analysis is considered exploratory and no primary conclusions about the efficacy of either HCL or verapamil will be based solely on the results of this analysis. If the interaction term is significant, separate results also will be reported (described below).
- In cohort A, the same constrained longitudinal analysis model described above for the primary analysis of C-peptide AUC at 52 weeks (Section 7.2) will be fit with the addition of a device by drug interaction. If there is evidence for an interaction at 52 weeks (p<0.05), the following additional analyses will be performed:
  - Baseline Characteristics
- A separate table for Cohort A, one column for each of the 4 combinations of HCL and Verapamil.
- HCL vs. non-HCL

- Summary statistics for C-peptide AUC at 52 weeks will be given separately for each of the 4 treatment group combinations. Boxplots will be given for baseline, 6, 13, 26, 39 and 52 weeks with one box for each of the 4 treatment combinations at each visit. The point estimate, 95% confidence interval and p-value at 52 weeks will be given from the model described above for the HCL effect separately in the verapamil and placebo groups. The HCL effect will also be estimated separately in cohort B.
  - Verapamil vs. Placebo
- Analogous analyses will be performed as described in the previous bullet reversing the roles of HCL and verapamil (Cohort A only).

### 10. Sensitivity Analyses

### 10.1 Confounding

420

423

424

432

433

437

441

443 444

445

- Imbalances between groups in important covariates are not expected to be of sufficient
- 426 magnitude to produce confounding. The primary analysis described above in Section 7 includes
- a fixed, pre-specified list of covariates. As an additional sensitivity analysis, any baseline
- demographic or clinical characteristics (see Section 14 below) observed to be imbalanced
- between HCL or verapamil treatment groups will be added as covariates in the primary analyses.
- The determination of a meaningful balance will be based on clinical judgement and not a p-
- value. This assessment of baseline differences will be made blinded to the outcome data.

# 10.2 Missing Data

- It is worth emphasizing that any statistical method for handling missing data makes a number of untestable assumptions. The goal will be to minimize the amount of missing data in this study so that results and conclusions will not be sensitive to which statistical method is used.
- To that end, a number of methods will be handle any missing data. As noted above in Section 7, the primary analysis will use the method of direct likelihood. Additional sensitivity analyses will handle missing data by:
  - Rubin's multiple imputation
- Multiple imputation with a pattern mixture model
  - Available cases only

### 11. Subgroup Analyses

- Subgroup analyses will be conducted separately for the two primary analyses (HCL and
- verapamil). Interpretation of the analyses will be made with caution and tests only performed if
- the overall treatment effect from the corresponding primary hypothesis is significant (P<0.05).
- The general approach for these exploratory analyses will be to add an interaction term for the
- subgroup factor by treatment into the model used for the primary analyses. A similar analysis
- will be repeated for time in range 70-180 mg/dL. The following baseline factors will be tested:
- Age (<12, ≥12 years old)

| 453<br>454 | <ul><li>Sex</li><li>Tanner staging (I vs II-V)</li></ul> |
|---|---|
| 454<br>455 | <ul> <li>Tanner staging (1 vs 11-v)</li> <li>Time since diagnosis at randomization</li> </ul> |
| 456 | <ul> <li>Presence of DKA at diagnosis at randomization</li> </ul> |
| 457 | HbA1c at randomization |
| 458 | C-Peptide AUC at randomization |
| 459 | Antibody levels at screening |
| 460 | Pre-existing autoimmune diseases |
| 461 | |
| 462 | The p-value for any categorical variable will only be calculated if there are a minimum of 10 |
| 463 | subjects per treatment group. |
| 464 | |
| 465 | 12. Additional Exploratory Analyses |
| 466 | 12.1 C-peptide |
| 467 | The following tabulations will be performed at 13, 26, 39, and 52 weeks by treatment group: |
| 468 | Peak C-peptide during a 2-hour MMTT |
| 469 | <ul> <li>Percentage of patients with peak C-peptide ≥ 0.2 pmol/ml</li> </ul> |
| 470 | |
| 471 | 12.2 HbA1c |
| 472 | The percent of participants with HbA1c < 6.5% and percent < 7.0% will be tabulated at 13, 26, 39, |
| 473 | and 52 weeks by treatment group. |
| 474 | |
| 475 | 12.3 CGM Metrics |
| 476 | For daytime and nighttime, each CGM metric listed in Section 5 will be tabulated accordingly at |
| 477 | 6, 13, 26, 39, and 52 weeks by treatment group. |
| 478 | |
| 479 | 12.4 Insulin |
| 480 | The following tabulations will be performed at 6, 13, 26, 39, and 52 weeks by treatment group: |
| 481 | Total daily insulin dose per kg |
| 482 | Basal:Bolus ratio |

484 12.5 C-peptide and Glycemic Control

483

488

To evaluate the relationship between C-peptide and glycemic control, scatterplots will be created at each time of the following factors on the horizontal axis, with C-peptide AUC on the vertical axis:

• CGM-measured % in range 70-180 mg/dL

- CGM-measured % above 180 mg/dL
- CGM-measured % below 70 mg/dL
- CGM-measured % below 54 mg/dL
- 492 Glucose CV

495 496

502

503

504

505

506 507

508

509

510

511

512

513 514

515

517

518

519

520

521

522 523

- 493 Mean HbA1c
  - HbA1c CV
    - Insulin dose adjusted percent time in range (70-180 mg/dL)

A longitudinal regression model will be fit with C-peptide as the dependent variable and time in range as the predictor variable separately for the HCL and non-HCL arms pooled over verapamil arms. Curves will be constructed for HCL and non-CL analogous to the DCCT analysis of HbA1c and retinopathy [5]. Similar curves will be constructed for verapamil and placebo arms and all four combinations if interaction is detected (see Section 9 above).

Similar to the model described above, a longitudinal regression model will be used to compare C-peptide between those who achieved high (> 85%) vs lower (< 65%) time in range separately for the HCL and non-HCL arms pooled over verapamil arms. The cutoffs for the high and low time in range groups may be adjusted after reviewing the distribution.

Additional exploratory analyses will be done using the other CGM metrics (and HbA1c) listed above and various combinations thereof. Model selection techniques with shrinkage (e.g., LASSO) will be used to determine the combination of CGM metrics that best predict C-peptide, potentially adjusting for confounding factors such as age and sex. Since these are exploratory analyses, the statistical methods used may be data-driven depending on results observed from initial analyses.

### 13. Safety Analyses

All reported adverse events will be sorted by date and listed.

For SH events, DKA events, and serious adverse events (excluding DKA and SH events), appropriate summary statistics for the following outcomes will be tabulated by treatment group.:

- Number of events per participant
- Number of participants with at least one event
- Incidence rate per 100 person-years

As described above for the efficacy analyses, safety comparisons of HCL versus non-HCL will combine cohorts A and B, and comparisons of verapamil versus placebo will be restricted to cohort A. Formal statistical comparisons will only be performed if at least 5 events occur during the study. The proportion of participants with at least one event will be compared using generalized estimating equations (GEE) logistic regression adjusting for age, and time from diagnosis to randomization. Clinical site will be treated as a repeated factor using a compound symmetry covariance structure. A risk-adjusted difference and 95% confidence interval for the

| 531 | percentages will | be calculated | l using the | method of Kleinman | and Norton | (4) | . If the mode | l does |
|---|---|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|---|---|

- not converge then Barnard's test will be used instead. Incidence rates will be compared using a
- Poisson regression model adjusting for age and time from diagnosis to randomization as fixed
- effects and clinical site as a random effect. Models for DKA outcomes will also include presence
- or absence of DKA at diagnosis as a covariate.
- For SH events, separate analyses also will be done for the outcomes listed above that will only
- include events that resulted in seizure or a loss of consciousness (if there are at least 5 such
- 538 events).
- For the verapamil vs. placebo comparison the frequency of adverse events stratified by MeDRA
- 540 class will be reported.

542

#### 14. Protocol Adherence and Retention

- Tabulations and figures by treatment group to assess protocol adherence will include:
- Flowchart accounting for all subjects according to treatment group for all visits
- Visit completion rates for each follow up visit
- Protocol deviations
  - Numbers and reasons for unscheduled visits and phone calls

547 548

HCL system use, verapamil, and placebo adherence will be tabulated at each time point and reported in a table.

551

552

### 15. Baseline Descriptive Statistics

- Baseline demographic, outcome, and covariate characteristics will be summarized with counts
- 554 (percentages), mean (SD), median (quartiles) as appropriate to the distribution. There will be two
- tables, one for HCL vs. non-HCL in the combined A+B cohort, and another for verapamil vs.
- Placebo, including only cohort A. For each of these tables, there will be a total column.
- 557 Age
- 558 Gender
- 559 Race
- 560 Ethnicity
- Annual Household income
- 562 Education
- 563 Health Insurance
- DKA at diagnosis
- 565 HbA1c lab
- 566 C-peptide AUC
- Time since diagnosis at randomization
- Tanner Staging (I vs II-V)

• Blood pressure (systolic/diastolic) 569 570 BMI 571 16. Device Issues 572 All reportable device issues occurring during the study will be tabulated and reported in a table. 573 574 575 17. Planned Interim Analyses No formal interim analyses or stopping guidelines are planned for this study. 576 577 The DSMB will review data for safety per the DSMB Standard Operating Procedures approximately every six months. The data to be reviewed will include information regarding 578 adverse events, device issues, and protocol adherence/deviations as they may relate to participant 579 safetv. 580 581 582 18. Multiple Comparisons 583 For the primary analyses, no adjustments for multiplicity will be made because two different 584 interventions are being tested separately. 585 For secondary analyses the false discovery rate (FDR) will be controlled using the adaptive 586 Benjamini-Hochberg procedure separately for the HCL and verapamil analyses. For these 587 analyses, the adjusted p-value and 95% confidence interval will be reported. 588 There will be no adjustments for multiple comparisons on safety analyses, sensitivity analyses, 589 or per protocol analyses. 590 591 592

### 18. References

- 1. Lachin JM, McGee PL, Greenbaum CJ, et al. Sample size requirements for studies of 593
- treatment effects on beta-cell function in newly diagnosed type 1 diabetes. PLoS One. 594
- 2011;6(11):e26471. 595
- 2. Ovalle F, Grimes T, Xu G, et al. Verapamil and beta cell function in adults with recent-onset 596
- type 1 diabetes. Nature medicine. 2018;24(8):1108-1112. 597
- 3. Greenbaum CJ, Beam CA, Boulware D, et al. Fall in C-Peptide during first 2 years from 598
- diagnosis: evidence of at least two distinct phases from composite type 1 diabetes TrialNet data. 599
- Diabetes 2012; 61(8): 2066-2073. 600

- 4. Kleinman LC, Norton EC. What's the risk? A simple approach for estimating adjusted risk
- measures from nonlinear models with logistic regression. Health Services Research 2009; 44(1):
- 603 2009 Feb.
- 5. Diabetes Control and Complications Trial Research Group: The relationship of glycemic
- exposure (HbA1c) to the risk of development and progression of retinopathy in the Diabetes
- 606 Control and Complications Trial. Diabetes, 1995; 44:968-983.